CLINICAL TRIAL: NCT01997996
Title: ProViS (Prolift+M TM and Vita Sexualis) Study
Brief Title: ProViS (Prolift+M and Vita Sexualis) Study
Acronym: ProViS
Status: Completed | Type: Observational
Sponsor: Dr. med. Tanja Hülder (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Tanja Hülder, Dr. med. Tanja Hülder, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: CTU 10/038
Record Dates: First submitted 2013-10-29; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; PROLIFT+M; Vita sexualis
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PROLIFT+M: Patients that undergo surgery due to prolapse POP ≥ stage II with PROLIFT+M device having had ≥ 2x/4 weeks sexual intercourse before surgery.

SUMMARY:
Transvaginal meshes (TVM) are indicated for the treatment of pelvic organ prolapse (POP) where surgical intervention is necessary. Due to a potential risk of de novo dyspareunia, TVM are mainly used in postmenopausal women and in case of recurrent POP. PROLIFT+M (Trademark) is based on a highly flexible material which is partially absorbable. We suggest that PROLIFT+M has less impact on the vita sexualis than conventional TVM and could also be used for the treatment of younger and/or sexually active women. This study observes women who are routinely treated with PROLIFT+M with regard to their sexual function before and after the surgery. The hypothesis is that there is no worsening in vita sexualis with PROLIFT+M.

ELIGIBILITY:
Inclusion Criteria:

* The patient understands the nature and content of the trial
* POP ≥ stage II (according to the POP-Q system (18))
* Sexual intercourse ≥ 2x/4 weeks
* Written informed consent
* Negative pregnancy test in women of childbearing potential
* Women ≥ 18 years

Exclusion Criteria:

* Concomitant surgery at the inner genitalis (e.g. colporrhaphy, sacrocolpopexy, sacrospinous fixation, hysterectomy); concomitant suburethral slings and bulking agents are allowed
* Unable to read or speak German
* Women < 18 years
* Women who are pregnant or breastfeeding or planning future pregnancies
* Acute infection(s), e.g. untreated urogenital infections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting specialist in hospitals and specialized doctor's offices scheduled to undergo Prolapse surgery.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
vita sexualis | 7 to 1 day Preoperative vs. 12 months (+/- 1 month) Postoperative
  No worsening in vita sexualis (decrease in total score Female Sexual Function Index (FSFI-d) of ≤ 3.3; max. score = 36) measured at 12 months (+/- 1 month) postoperatively as compared to the preoperative score.

SECONDARY OUTCOMES:
pain during sexual intercourse | 7 to 1 day Preoperative vs. 12 months (+/- 1 month) Postoperative
  No worsening in pain during sexual intercourse (decrease in weighted pain subscore FSFI-d of ≤ 1; max score = 6) measured at 12 months (+/- 1 month) postoperatively compared to preoperative.
Assessment of pelvic floor function | 7 to 1 day Preoperative vs. 12 months (+/- 1 month) Postoperative
  Assessment of pelvic floor function using the validated German pelvic floor questionnaire at 12 months (+/- 1 month) postoperatively compared to preoperative (Deutscher Beckenboden-Fragebogen, validated German Version of the Australian Pelvic Floor Questionnaire
Assessment of patient satisfaction | 12 months (+/- 1 month) Postoperative
  Assessment of patient satisfaction at 12 months (+/- 1 month) postoperatively using the visual analogue scale (VAS), question regarding reoperation and patient global (PGI) question.VAS: On top of two scales, the question "How satisfied are you with the result of your operation?" is placed. (Facial expressions are put above the line to express satisfaction visually). In addition, the following two questions are asked: "Would you have the operation done again?" and "In the past 12 months how would you rate your condition as opposed to before your recent pelvic floor operation: much better/a little better/about the same/a little worse/much worse" (PGI question).
Assessment of recurrent POP (POP-Q ≥ stage II) | 3 months (12 weeks +/- 2) and 12 months (+/- 1 month) postoperatively
  Assessment of recurrent POP (POP-Q ≥ stage II in the operated compartment(s)), mesh erosion/exposure; each measured 3 (12 +/- 2 weeks) and 12 months (+/- 1 month) postoperatively by clinical examination (Speculum, palpation, POP-Q)
Safety | until 12 months (+/- 1 month) postoperatively
  Safety (documentation and assessment of medical device incidents; serious incidents and near incidents will be reported to the competent authorities)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Hülder, Dr.med., Study Chair — Cantonal Hospital of St. Gallen
Locations (4):
- Germany (3):
  - Klinikum Augsburg, Augsburg, Bavaria
  - Universitätsklinikum des Saarlandes, Homburg/Saar, Saarland
  - DRK Krankenhaus Chemnitz-Rabenstein, Chemnitz, Saxony
- Kantonsspital St.Gallen, Sankt Gallen, St.Gallen, Switzerland